CLINICAL TRIAL: NCT03801005
Title: Immunophenotyping of Blast Cells and Immune Effector Cells in Peripheral Whole Blood and Bone Marrow Samples From AML and MDS Patients
Brief Title: Immunophenotyping of Blast Cells and Immune Effector Cells in Peripheral Whole Blood and Bone Marrow Samples From AML and MDS Patients (AML)
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-43
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood and Marrow sample — Twenty patients will be included in a prospective way over a period of nine months. No additional medullary or serum samples will be carried out in addition to those required for the clinical routine. Only an additional blood sample taken during a routine blood test will be recovered as part of the research. Just as some leftover bone marrow, taken as part of a usual unused follow-up will be recovered as part of this trial.
  The persons concerned will be recruited on the occasion of their hospitalisation in one of the hematology services participating in the research, or during their consultation with one of the hematologists of the corresponding service (or services). On this occasion, detailed information on their pathology and research will be given, as well as the information document on the proposed research protocol.

SUMMARY:
The objective of this study is to evaluate the immune profile of blast cells and immune effector cells in paired peripheral whole blood and bone marrow samples from AML and MDS patients by standardized flow cytometry. A special emphasis will be focused on monitoring expression of CD200 as well as PGP-170 (MDR1) on blasts cells.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* No pregnant woman
* Patient with myelodysplastic syndrome (with excess blasts) or acute myeloid leukemia
* Presence of a monitored serum blastose
* Patient who can obtain free and informed consent (speaks French, no guardianship or curatorship)

Exclusion Criteria:

* Minor Patient (< 18 years old)
* Medical or psychological Condition that could interact with the ability to understand the study,
* Pregnant or lactating women,
* Major persons under guardianship or under the protection of justice
* Persons deprived of their liberty by a judicial or administrative decision
* Lack of information and opposition to its participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with myelodysplastic syndrome (with excess blasts) or acute myeloid leukemia
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
evaluate the immune profile of blast cells and immune effector cells in paired peripheral whole blood and bone marrow samples from AML and MDS patients by standardized flow cytometry. | 9 mounths

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique - Hopitaux de Marseille, Marseille, France